CLINICAL TRIAL: NCT02776800
Title: A Randomized, Controlled Study of Allevyn Life in the Management of Wounds in Home Health Care
Brief Title: Managing Wounds With Allevyn Life in a Home Health Care Environment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business Decision
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CE054ALF
Record Dates: First submitted 2016-05-16; First posted 2016-05-18 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Wounds and Injuries
Keywords: Wound; Surgical Wound; Trauma Wound; Home Health Care; Home Health Nurse; Pressure Ulcer; Diabetic Foot Ulcer; Venous Leg Ulcer; Arterial Ulcer; Wound Dehiscence; Open Wound
MeSH Terms: conditions — Wounds and Injuries; Surgical Wound; Pressure Ulcer; Diabetic Foot; Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allevyn Life (Experimental): Foam Dressing
  Interventions: Device: Allevyn Life
- Foam Dressing (Other): Standard Care - Foam Dressing
  Interventions: Device: Foam dressing with an integrated adhesive border

INTERVENTIONS:
Device: Allevyn Life
  Arms: Allevyn Life
Device: Foam dressing with an integrated adhesive border — Foam dressing normally used by the home health agency
  Arms: Foam Dressing

SUMMARY:
When elderly patients need help caring for wounds, physicians may refer patients to home health care providers. The home health provider sees the patient in the patient's home and assists the patient with wound care. Working with the patient's physician, the home health provider will use the appropriate wound covering ("dressing" or "bandage") to cover the wound. The goal of the home health provider is to ensure that the wound stays clean and progresses toward closure. The home health provider will conduct in-home patient visits at appropriate intervals to assess the status of the wound.

Extensive resources are required to see patients in their own homes. If a dressing could effectively manage wounds and allow longer time between in-home visits (without affecting patient safety or progress of the wound toward closure), then resources could be saved. Thus, newer dressings are designed for longer wear times, using advanced foam pads and adhesives that help keep the dressing in place. The hypothesis of this study is that the use of Allevyn Life will decrease the number of in-home visits by home health providers without sacrificing patient safety.

ELIGIBILITY:
INCLUSION CRITERIA

1. The informed consent document must be read, signed, and dated by the subject or the subject's legally authorized representative before conducting any study procedures or exams. 2. Subjects sixty-five (65) years of age or older. Subjects may be of either sex and of any race.

3. Willing and able to allow home health clinician to conduct all required study visits.

4. The subject (or caregiver) must be able to follow instructions, including the ability to have regular contact with the home health clinician between study visits.

5. Are covered by traditional Medicare. 6. Have a wound that is suitable for treatment with a foam dressing and can be appropriately covered by a single piece of ALLEVYN Life or the comparator dressing.

7. At Screening, wound exudate must be moderate to heavy, as determined by the home health clinician.

8. Target wound may be a trauma wound, chronic wound, or post-surgical wound. 9. Wound care is the primary reason for the home health clinician visits and determines the frequency of home health visits. Subjects may have other comorbidities, but these cannot be the determining factor in scheduling the frequency of the home health visits.

EXCLUSION CRITERIA

1. Contraindications or hypersensitivity to the use of the study dressings or their components (e.g., adhesive)
2. Any wound that requires an additional covering (e.g., compression dressing, cast, etc.) over the study dressing that prevents daily visualization of the dressing under study.
3. Target wound that requires daily dressing changes due to topical wound treatment (e.g., daily applications of ointments, creams, etc.)
4. Target wound and dressing that cannot be visualized by the subject or subject's caregiver.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08 (Estimated); Primary Completion 2017-07 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Number of home health clinician visits in each group | 60 days

SECONDARY OUTCOMES:
Home health provider time on-site | 60 days
Total cost of each treatment group | 60 days
Number of visits required compared to number initially anticipated | 60 days
Assess the Cardiff Wound Impact Schedule | 60 days
Average dressing wear time | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Smith & Nephew, Inc.; Jaime E Dickerson, PhD, Study Director — Smith & Nephew, Inc.
Locations (3):
- United States (3):
  - Tustin, California
  - Wichita, Kansas
  - McAllen, Texas

IPD SHARING:
Plan to Share IPD: No